CLINICAL TRIAL: NCT03528525
Title: Beijing Children's Hospital
Brief Title: Registry Study on Respiratory Monogenic Diseases in Chinese Children
Status: Recruiting | Type: Observational
Sponsor: Kunling Shen (Other)
Collaborators: Capital Institute of Pediatrics, China (Other); Shengjing Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Children's Hospital of Chongqing Medical University (Other); The first clinical college of Guangzhou medical university (Unknown); Guangzhou Women and Children's Medical Center (Other); Yuying Children's Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Kunling Shen, Beijing Children's Hospital, Beijing Children's Hospital
Organization: Beijing Children's Hospital (Other)
Other Study IDs: BCHlung 010
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Monogenic Diseases
Keywords: Diseases; Children; Respiratory; Monogenic diseases; China
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Monogenic diseases cases

INTERVENTIONS:
Other:  — observation

SUMMARY:
This study is a multicenter, prospective cohort study of patients diagnosed with respiratory monogenic diseases, the clinical information of recruited patients, including clinical manifestations, lung function, chest imaging, quality of life and other indicators, will be followed for 5 years.

DETAILED DESCRIPTION:
All new cases of respiratory monogenic diseases was confirmed or diagnosed at each center from the beginning of the study are made the investigation of the clinical manifestations and specific tests by the standard diagnostic process.Then all the patients' following clinical data will be followed for 5 years: clinical manifestations, lung function, chest imaging (once per year), gene test, quality of life and other indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 0-18 years, male and female.
2. Any organ system symptoms consistent with the diagnostic points of respiratory monogenic diseases.
3. Agree to retain specimens related to disease research and agree to store the specimens in the sample bank.
4. willing and able to cooperate with long-term follow-up.
5. The guardian of the child has a full understanding of the purpose of the study, a basic understanding of the clinical research program, and voluntarily allows the child to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. It is unable to provide complete medical records or the current condition can not accept the diagnosis process
2. She or he cannot agree to participate in the study.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who was confirmed diagnosis as respiratory monogenic diseases at the certain hospitals (sponsor and collaborators)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lung function on the spirometry | 1 year later
  forced expiratory volume at one second (FEV1) in Liter

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's hospital, Beijing, Beijing Municipality, China